CLINICAL TRIAL: NCT01230320
Title: Simplified vs. Conventional Methods for the Fabrication of Complete Dentures in a Public Health Setting
Brief Title: Simplified vs. Conventional Methods for Complete Denture Fabrication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Raphael Freitas de Souza, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FORP-PT-001; 2010.1.971.58.0 (Other: Institutional Review Board (FORP-USP)); 2010/09381-9 (Other Grant/Funding Number: FAPESP (São Paulo Research Foundation))
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: Cost estimates; Complete Denture; Dental Economics; Dental Impression Technique; Denture Retention; Edentulous; Edentulism; Oral Health-Related Quality of Life; Patient Acceptance of Health Care; Patient Satisfaction; Quality of Health Care; Quality of Life
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simplified (S) technique (Experimental): Complete dentures fabricated according to a simplified technique, divided into the following four sessions:
  1. Maxillary and mandibular casts will be obtained from irreversible hydrocolloid impressions made in stock trays.
  2. Record bases will be adjusted according to vertical dimension and centric relation measurements, without facebow transfer. Casts will be mounted in a semi-adjustable articulator using standardized measures and artificial teeth will be selected.
  3. Trial dentures will be evaluated for esthetics and maxillomandibular relationships.
  4. Insertion of finished dentures.
  Interventions: Procedure: Denture fabrication technique
- Conventional (C) technique (Active Comparator): Complete dentures fabricated according to a conventional technique:
  1. Initial impression and the obtainment of custom trays;
  2. Final impression with border molding using compound;
  3. Facebow transfer;
  4. Determination of maxillomandibular relationship;
  5. Try-in of anterior teeth;
  6. Try-in of posterior teeth;
  7. Insertion of finished dentures.
  Interventions: Procedure: Denture fabrication technique

INTERVENTIONS:
Procedure: Denture fabrication technique — Sequence of procedures involved with the fabrication of conventional complete dentures. Examples of common procedures are:
  1. the reproduction of denture-bearing tissues by means of impression techniques and casts;
  2. the registration of maxillo-mandibular relations;
  3. try-in of artificial teeth and carved denture bases.
  Other Names: - Fabrication of complete dentures;; - Complete denture fabrication technique.

SUMMARY:
BACKGROUND: The fabrication of complete dentures traditionally involves a series of complex technical procedures. Those procedures include two impressions for each jaw, the registration of the relationship between the upper teeth and the patient's head and usually two appointments for tooth try-in. However, recent studies have questioned the real need for such complex procedures. Simplified methods could have similar results if compared with conventional ones, and dentures would be delivered faster and with lower costs.

OBJECTIVES: This study aims to compare the effectiveness complete dentures fabricated with a simplified or conventional method.

METHODS: Eighty edentulous patients who requested treatment by maxillary and mandibular complete denture in a public dental clinic inside the University of Sao Paulo - Ribeirão Preto Dental School will be randomly divided into two groups. Group S will receive new dentures fabricated by a simplified method, whereas Group C will received new dentures according to a conventional method. Participants will complete a questionnaire for denture satisfaction and the oral health-related quality of life, 3 and 6 months after treatment. At the same time, a specialist in dental prostheses will evaluate the quality of new dentures.

DETAILED DESCRIPTION:
Complete edentulism can be considered as an important public health problem, particularly in the elderly. The prevalence of edentulism among adults aged 65 or more years is still high in several countries, such as Canada (58%), Saudi Arabia (31-46%), United Kingdom (46%), China (11%) and India (19%). Normative needs of maxillary and mandibular complete dentures in Brazilian elders were estimated to be 16% and 24%, respectively. This way, the epidemiologic aspect reinforces the need for cost-effective methods when treating patients with complete dentures.

The conventional methods for fabrication of complete dentures demand a comprehensive sequence of clinical and laboratorial procedures. Those methods seem to be accepted and taught by most of the American and Brazilian dental schools. However, it has been argued whether they are necessary for the obtainment of adequate dentures. Several approaches were described in attempt to simplify clinical and laboratorial stages, i.e. the fabrication of denture bases directly on casts obtained from irreversible hydrocolloid impressions made in stock trays. Other simplified approaches include the fabrication without facebow transfer, alternative occlusal schemes (i.e. lingualized occlusion) and duplication techniques.

A few recent randomized clinical trials have provided some high level evidence about the efficacy of simplified methods. We ran the following search strategy for PubMed at October 2010:

(overdenture or ((removable or complete) and denture)) and ((techni* or fabricat* or simpl* or tradition*) or (impression* or occlus* or (facebow or face-bow) or remount* or adjust*)) and (((randomized controlled trial [pt]) OR (controlled clinical trial [pt]) OR (randomized [tiab]) OR (placebo [tiab]) OR (drug therapy [sh]) OR (randomly [tiab]) OR (trial [tiab]) OR (groups [tiab])) AND (humans [mh]))

After reading the 470 titles and abstracts, and examining possible reports of randomized clinical trials, only two studies that attempted to evaluate simplified methods for denture fabrication were found.

One of the studies compared a simplified and a conventional method for complete denture fabrication by a parallel arms trial. The difference between the methods was the use of a second impression, facebow transfer and remount by the conventional approach. No significant difference between the groups was found for the outcome variables tested - denture quality and patient satisfaction. The other trial compared the relative efficacy of complete dentures fabricated according to two occlusal concepts, by means of a crossover design. A more complex method employed a facebow transfer with recordings of condylar inclination, gothic arch tracing and bilateral balanced occlusion. The simplified technique used no facebow transfer, manual technique for the record of centric occlusion and canine guidance. Denture satisfaction was not influenced by the fabrication method.

The current evidence raises doubt about the relevance of some procedures involved in the fabrication of complete dentures. Despite the high quality of the previously cited trials, further studies could use a more pragmatically approach such as testing methods in public health patients. Moreover, data from additional studies could be summarized in the future by means of meta-analysis and thus evidence would be stronger. In summary, such studies may provide support to either:

1. Improve access of the edentulous patients to complete denture treatment by lowering costs and complexity;
2. Reinforce the importance of technical procedures during denture fabrication.

OBJECTIVES

To compare complete dentures fabricated with a simplified technique and conventional prostheses for the rehabilitation of edentulous patients, after 3 and 6 months of wearing.

The null hypothesis will be that mean values of oral health-related quality of life for pairs of dentures fabricated by the simplified and the conventional dentures are similar. Similar secondary hypotheses will be considered for the secondary variables.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous for at least 1 year
* Patients requesting new maxillary and mandibular complete dentures
* Mental receptiveness
* Good understanding of spoken Portuguese

Exclusion Criteria:

* Debilitating systemic diseases
* Pathologic changes of residual edentulous ridges
* Dysfunctional disorders of the masticatory system

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life | 6 months
  To be assessed by means of the Brazilian version of the OHIP-EDENT.

SECONDARY OUTCOMES:
Denture satisfaction | 6 months
  To be assessed by specific questionnaires.
Denture quality | 3 months
  To be assessed by means of clinical exam following a specific form.
Post-insertion adjustments | 14 days
  Necessary post-insertion, as done routinely for conventional denture patients.
Treatment costs | 6 months
  This outcome will be measured by means of specific forms, according to 2 components:
  * Direct costs: cost of labor, materials, radiographs and medications;
  * Indirect costs: patient's time and transportation expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael F de Souza, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Ribeirão Preto Dental School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Institutional page of the Ribeirão Preto Dental School (research site) — http://www.forp.usp.br
- See also: Principal Investigator´s CV — http://sistemas3.usp.br/tycho/CurriculoLattesMostrar?codpub=F7A61880194F